## Investigating Compassion-Based Guided Self-Help for Depression in People with Skin Conditions

Elaine Clarke

NCT04132973

Informed consent form

Document date: 15<sup>th</sup> Nov 2019

Uploaded to PRS: 19<sup>th</sup> Aug 2021

Research Study: An Acceptability and Feasibility Study of a Compassion-Based Guided Self-Help Intervention for Depression in People with Skin Conditions

## Appendix B Consent statement

| | Agree | Disagree |
|---|---|---|
| I confirm that I am over the age of 18 and that I have been diagnosed with a skin condition by a medical professional. | О | О |
| I have read and understood the participant information sheet<br>and have had the opportunity to ask questions of the researcher<br>by email. | О | 0 |
| I understand that taking part in this study will involve answering questions about my mental health and skin condition and carrying out activities that may increase my awareness of preexisting psychological distress. | 0 | O |
| I understand that my participation in this study is voluntary and that I may withdraw from the study at any time, without giving a reason and without any adverse consequences. | O | 0 |
| I am aware that this study will be administered online and that I will be contacted regularly by email during the study period, but that my personal details will not be disclosed to any third parties nor will I be identified or identifiable in any of the results. | О | O |

15/11/2019 viii